CLINICAL TRIAL: NCT03110757
Title: A Phase Ib Study of the Safety, Reactogenicity, and Immunogenicity of Sm-TSP-2/Alhydrogel(R) With or Without AP 10-701 for Intestinal Schistosomiasis in Healthy Exposed Adults
Brief Title: A Phase Ib Study of the Safety, Reactogenicity, and Immunogenicity of Sm-TSP-2/Alhydrogel)(R) With or Without AP 10-701 for Intestinal Schistosomiasis in Healthy Exposed Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 14-0100; HHSN272201300015I
Record Dates: First submitted 2017-03-21; First posted 2017-04-12 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01-26

CONDITIONS: Schistosomiasis
Keywords: AP 10-701; healthy adults; Immunogenicity; Phase Ib; Reactogenicity; Safety; Schistosomiasis; Sm-TSP-2/Alhydrogel®
MeSH Terms: conditions — Schistosomiasis | interventions — GLA-AF adjuvant; Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group A (Experimental): 10mcg Sm-TSP-2/Alhydrogel® (n=8)
  Interventions: Biological: Sm-TSP-2/Alhydrogel
- Group B (Experimental): 10mcg Sm-TSP-2/Alhydrogel®/+ AP 10-701 (n=8)
  Interventions: Biological: GLA-AF; Biological: Sm-TSP-2/Alhydrogel
- Group D (Experimental): 30mcg Sm-TSP-2/Alhydrogel® (n=8)
  Interventions: Biological: Sm-TSP-2/Alhydrogel
- Group E (Experimental): 30mcg Sm-TSP-2/Alhydrogel®/+ AP 10-701 (n=8)
  Interventions: Biological: GLA-AF; Biological: Sm-TSP-2/Alhydrogel
- Group G (Experimental): 100mcg Sm-TSP-2/Alhydrogel® (n=8)
  Interventions: Biological: Sm-TSP-2/Alhydrogel
- Group H (Experimental): 100mcg Sm-TSP-2/Alhydrogel®/+ AP 10-701 (n=8)
  Interventions: Biological: GLA-AF; Biological: Sm-TSP-2/Alhydrogel
- Pooled Active Comparator Group (Active Comparator): Euvax B Hepatitis B vaccine (n=12)
  Interventions: Biological: Hepatitis B Virus Vaccine (Recombinant)

INTERVENTIONS:
Biological: GLA-AF — Previously referred to as Gluco-pyranosylphospho-lipid A aqueous formulation (GLA-AF). It is a toll-like receptor-4 agonist
  Arms: Group B; Group E; Group H
Biological: Hepatitis B Virus Vaccine (Recombinant) — A non-infectious subunit viral vaccine derived from hepatitis B surface antigen (HBsAg) produced in yeast cells.
  Arms: Pooled Active Comparator Group
Biological: Sm-TSP-2/Alhydrogel — Sm-TSP-2/Alhydrogel
  Arms: Group A; Group B; Group D; Group E; Group G; Group H

SUMMARY:
The study will be conducted as a randomized, controlled, double blind Phase 1b dose-escalating clinical trial in up to 60 healthy adult males and non-pregnant females living in the S. mansoni-endemic area of Americaninhas, Brazil. The primary objective of this trial is to assess the safety and reactogenicity of ascending doses of Sm-TSP-2/Alhydrogel(R) (10mcg, 30mcg, or 100mcg) vaccine with or without AP 10-701 given as three doses administered on Days 1, 57, and 113.

DETAILED DESCRIPTION:
The study will be conducted as a randomized, controlled, double blind Phase 1b dose-escalating clinical trial in up to 60 healthy adult males and non-pregnant females living in the S. mansoni-endemic area of Americaninhas, Brazil. The study will recruit up to 60 healthy adult males and non-pregnant females to test two formulations of Sm-TSP-2 vaccine (adjuvanted with Alhydrogel(R) only, or with Alhydrogel(R) plus AP 10-701), each at 3 different doses of antigen: 10mcg, 30mcg, and 100mcg. The study will use a dose-escalation cohort design, in which escalation to the next dose cohort will be determined based on evaluation of pre-defined escalation criteria requiring 7 day safety data to be examined after all subjects in the current cohort have received their first dose of vaccine. Cohorts will be enrolled sequentially. For each Cohort (1-3), an initial 5 subjects (2 Sm-TSP-2/Alhydrogel(R), 2 Sm-TSP-2/Alhydrogel(R)/AP 10-701, and 1 Euvax B Hepatitis B vaccine) will be enrolled, randomized, vaccinated, and have completed Visit 02 (Day 2), before enrolling the rest of the cohort. As with dose-escalation decisions, evidence of significant reactogenicity will require further review prior to proceeding. The primary objective of this trial is to assess the safety and reactogenicity of ascending doses of Sm-TSP-2/Alhydrogel(R) (10mcg, 30mcg, or 100mcg) vaccine with or without AP 10-701 given as three doses administered on Days 1, 57, and 113. The secondary objectives used to evaluate the immunogenicity are: (1) to assess the IgG antibody response to Sm-TSP-2 using an indirect enzyme-linked immunosorbent assay (ELISA) at Day 127, (2) to assess the IgG antibody response to Sm-TSP-2 using an indirect ELISA at 14 days after dose one and two and Days 203, 293, and 478 (3, 6, and 12 months after the third dose) of Sm-TSP-2/Alhydrogel(R) (10mcg, 30mcg, or 100mcg) with or without AP 10-701, and (3) to assess the duration of the IgG antibody response to Sm-TSP-2 using an indirect ELISA following receipt of three doses of Sm-TSP-2/Alhydrogel(R) (10mcg, 30mcg, or 100mcg) with or without AP 10-701.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study procedures.
2. Able to understand and comply with planned study procedures and be available for all study visits.
3. Male or non-pregnant female aged 18 to 50, inclusive at the time of enrollment.
4. Are in good health, as determined by vital signs (oral temperature, pulse, and blood pressure), medical history, and brief physical examination at screening.

   -Existing medical diagnoses or conditions (except those in the Subject Exclusion Criteria) must be deemed as stable chronic medical conditions. A stable chronic medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last 3 months (90 days) and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months (180 days). Any change due to change of health care provider, or that is done for financial reasons, as long as in the same class of medication, will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a violation of this inclusion criterion. Subjects may be on chronic or as needed medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity. Topical, nasal, and inhaled medications (with the exception of corticosteroids as outlined in the Subjects Exclusion Criteria), vitamins, and contraceptives are permitted.
5. Vital signs (oral temperature, pulse, and blood pressure) are all within normal protocol-defined ranges.

   -The normal protocol-defined ranges for vital signs include (a) oral temperature less than 38.0 degrees celsius, (b) pulse 50 to 100 bpm, inclusive, (c) systolic blood pressure 85 to 150 mmHg, inclusive, and (d) diastolic blood pressure 55 to 90 mmHg, inclusive. Pulse rate <50 is acceptable for 2nd and 3rd vaccinations if the subject is otherwise healthy with documented sinus bradycardia at baseline.
6. Laboratory tests (alanine aminotransferase, creatinine, white blood cell count, hemoglobin, and platelets) are all within protocol-defined reference ranges.

   -The protocol-defined ranges for laboratory tests include (a) alanine aminotransferase (ALT) of less than 1.25-times the upper reference limit, (b) creatinine less than 1.25 times the upper reference limit (c) white blood cells (WBC) between 3.3 x10^3/uL and 10.4 x10^3/uL, inclusive, (d) hemoglobin 11.4 g/dL or greater for females or 12.1 g/dL or greater for males, (e) platelets greater than 130 x10^3/uL. Laboratory test results for 2nd and 3rd vaccinations may be at Grade 1 if considered unrelated to study product.
7. Urinalysis with no greater than trace protein and negative for glucose.
8. Female subjects of childbearing potential must agree to practice highly effective contraception for a minimum of 30 days prior to study product exposure and for 30 days after last vaccination.

   * Female subjects who are surgically sterile via tubal sterilization, bilateral oophorectomy or hysterectomy or who have been postmenopausal for greater than 1 year are not considered to be of childbearing potential.
   * Highly effective methods of contraception are defined as having low failure rates (i.e. less than 1% per year) when used consistently and correctly and may include, but are not limited to, abstinence from intercourse with a male partner, monogamous relationship with a vasectomized partner, male condoms or diaphragm with spermicide, intrauterine devices, and licensed hormonal methods.
9. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.
10. Able to correctly answer all questions on the informed consent comprehension questionnaire.

Exclusion Criteria:

1. Has the intention to become pregnant within 5 months after enrollment in this study.
2. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after their last study vaccination.
3. Has an acute illness, including a documented oral temperature of 38.0 degrees celsius or greater, within 72 hours prior to vaccination.
4. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
5. Is immunosuppressed as a result of an underlying illness or treatment.

   -Causes for immunosuppression may include, but are not limited to, poorly-controlled diabetes mellitus, cirrhosis, renal insufficiency, active neoplastic disease or a history of any hematologic malignancy, connective tissue disease, organ transplant.
6. Using or intends to continue using oral or parenteral steroids, high-dose inhaled steroids (>800 µg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
7. Positive hepatitis B surface antigen (HBsAg)
8. Positive confirmatory test for HIV infection
9. Positive confirmatory test for hepatitis C virus (HCV) infection
10. Volunteer has had a history of alcohol or illicit drug abuse during the past 24 months.
11. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
12. History of a severe allergic reaction or anaphylaxis to known components of the study vaccines.
13. Has an acute or chronic medical condition that, in the opinion of the investigator, would render participation in this study unsafe or would interfere with the evaluation of responses.

    -This includes, but is not limited to: known liver disease, renal disease, neurological disorders, visual field defects, cardiac disorders, pulmonary disorders, diabetes mellitus, and transplant recipients.
14. History of splenectomy
15. Is participating or plans to participate in another clinical trial with an interventional agent during the duration of the study.

    -This may include other licensed or unlicensed vaccines, drugs, biologics, devices, blood products, or medications.
16. Received any licensed live vaccine within 30 days or any licensed inactivated vaccine within 14 days prior to the first study vaccination.
17. Planned receipt of any vaccine from the first study vaccination through 28 days after the last study vaccination.
18. Has any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
19. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
20. Anti-Sm-TSP-2 IgE antibody level above ELISA reactivity threshold.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
The occurrence of new-onset chronic medical conditions (including AESI) | From Day 1 to Day 478
The occurrence of solicited injection site reactogenicity | From Day 1 to Day 7
The occurrence of solicited injection site reactogenicity | From Day 113 to Day 120
The occurrence of solicited injection site reactogenicity | From Day 57 to Day 64
The occurrence of solicited systemic reactogenicity | From Day 1 to Day 7
The occurrence of solicited systemic reactogenicity | From Day 113 to Day 120
The occurrence of solicited systemic reactogenicity | From Day 57 to Day 64
The occurrence of study vaccine-related SAEs | From Day 1 to Day 478
The occurrence of vaccine-related clinical safety laboratory adverse events | Day 113
The occurrence of vaccine-related clinical safety laboratory adverse events | Day 120
The occurrence of vaccine-related clinical safety laboratory adverse events | Day 57
The occurrence of vaccine-related clinical safety laboratory adverse events | Day 64
The occurrence of vaccine-related clinical safety laboratory adverse events | Day 8

SECONDARY OUTCOMES:
The anti-Sm-TSP-2 IgG antibody response using an indirect ELISA | Day 15
The anti-Sm-TSP-2 IgG antibody response using an indirect ELISA | Day 203
The anti-Sm-TSP-2 IgG antibody response using an indirect ELISA | Day 293
The anti-Sm-TSP-2 IgG antibody response using an indirect ELISA | Day 478
The anti-Sm-TSP-2 IgG antibody response using an indirect ELISA | Day 71
The anti-Sm-TSP-2 IgG level using an indirect ELISA | Day 127

CONTACTS AND LOCATIONS:
Locations (1):
- Americaninhas Vaccine Center, Novo Oriente, Minas Gerais, Brazil

REFERENCES:
- [Derived] Diemert DJ, Correa-Oliveira R, Fraga CG, Talles F, Silva MR, Patel SM, Galbiati S, Kennedy JK, Lundeen JS, Gazzinelli MF, Li G, Hoeweler L, Deye GA, Bottazzi ME, Hotez PJ, El Sahly HM, Keitel WA, Bethony J, Atmar RL. A randomized, controlled Phase 1b trial of the Sm-TSP-2 Vaccine for intestinal schistosomiasis in healthy Brazilian adults living in an endemic area. PLoS Negl Trop Dis. 2023 Mar 30;17(3):e0011236. doi: 10.1371/journal.pntd.0011236. eCollection 2023 Mar. PMID 36996185